CLINICAL TRIAL: NCT04063579
Title: Cardiac Magnetic Resonance Assessment for Heart Failure With Preserved Ejection Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UW18-022
Record Dates: First submitted 2019-08-16; First posted 2019-08-21 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — Echocardiography; Cardiac Catheterization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with heart failure with preserved ejection fraction (Experimental)
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance, Echocardiogram, Blood investigation (NT-proBNP), cardiac catheterization
- Non-heart failure patients (Experimental)
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance, Echocardiogram, Blood investigation (NT-proBNP), cardiac catheterization
- Normal Volunteers (Experimental)
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance, Echocardiogram, Blood investigation (NT-proBNP)

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic Resonance, Echocardiogram, Blood investigation (NT-proBNP), cardiac catheterization — Imaging, blood tests, LV pressure measurement
  Arms: Non-heart failure patients; Patients with heart failure with preserved ejection fraction
Diagnostic Test: Cardiac Magnetic Resonance, Echocardiogram, Blood investigation (NT-proBNP) — Imaging and Blood tests
  Arms: Normal Volunteers

SUMMARY:
This is a prospective study that aims to define the utility of cardiac magnetic resonance feature tracking (CMR-FT) as a non-invasive quantification tool to assess diastolic functionality in patients with Heart Failure with preserved ejection fraction.

DETAILED DESCRIPTION:
Despite the increasing prevalence and poor prognosis of HFpEF worldwide, it is facing diagnostic challenges due to its non-specific clinical manifestations. Currently, echocardiography serves as the main diagnostic tool, but alternatives are limited to less preferred invasive procedures in most clinical situations.

It is therefore proposed to investigate HFpEF using cardiovascular magnetic resonance imaging (CMR), as an alternative non-invasive diagnostic tool which carries lower risk than invasive procedures.

The study aims to: (1) access the utility of CMR-FT as a new indicator to diagnose diastolic dysfunction by differentiating HFpEF patients from non-HFpEF patient and normal volunteers. (2) Compare accuracy of CMR-FT to CMR tagging and phase contrast imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with symptoms and signs suggestive of HFpEF
* Patients undergoing coronary catheterisation for stable chest pain with no evidence of diastolic dysfunction, heart failure, infarct, left ventricular ejection fraction <50% or significant coronary artery disease (ie. >50% narrowing of one or more coronary arteries)
* Volunteers must be asymptomatic with no cardiac risk factors and no previous cardiac history

Exclusion Criteria:

* Patients suspected to have HFpEF but echocardiography and/or invasive pressure measurements do not confirm diagnosis of HFpEF.
* Significant underlying ischaemia based on clinical history and non-invasive imaging or catheter coronary angiography if indicated.
* Contraindication to CMR study
* Estimated glomerular filtration rate <30 ml/min/1.73 m2
* More than moderate valvular disease
* Severe pulmonary disease (ie. FEV1 <- 50% predicted)
* Cardiomyopathy
* Constrictive pericarditis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of feature tracking diastolic strain rate to diagnose diastolic dysfunction by differentiating HFpEF patients from the non-HFpEF patients and normal volunteers | 2 years

SECONDARY OUTCOMES:
Complication rate of cardiac catheterisation | 2 years
Unexpected findings by CMR (eg. Cardiac amyloidosis) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Result] Ng MY, Kwan CT, Yap PM, Fung SY, Tang HS, Tse WWV, Kwan CNF, Chow YHP, Yiu NC, Lee YP, Fong AHT, Hwang S, Fong ZFW, Ren QW, Wu MZ, Wan EYF, Lee KCK, Leung CY, Li A, Montero D, Vardhanabhuti V, Hai J, Siu CW, Tse HF, Pennell DJ, Mohiaddin R, Senior R, Yiu KH. Diagnostic accuracy of cardiovascular magnetic resonance strain analysis and atrial size to identify heart failure with preserved ejection fraction. Eur Heart J Open. 2023 Mar 7;3(2):oead021. doi: 10.1093/ehjopen/oead021. eCollection 2023 Mar. PMID 36992915